CLINICAL TRIAL: NCT07248904
Title: The Effect of a Transtheoretical Model-Based Educational Intervention on First-Year Nursing Students' HPV Knowledge, Health Beliefs, and Vaccination Behavior Intentions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, MÜJDE KERKEZ, Asist. Prof. Dr., Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTM-HPV-001
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus (HPV); Papillomavirus Vaccines; Health Knowledge, Attitudes, Practice; Students, Nursing; Health Behavior
MeSH Terms: conditions — Behavior; Health Behavior

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group randomized controlled design. Participants are first-year nursing students who will be randomly assigned, using simple randomization, to either the intervention group or the control group. The intervention group will receive a Transtheoretical Model (TTM)-based structured educational program tailored to the participant's stage of readiness for HPV vaccination. The control group will receive no structured education during the study period. Both groups will complete baseline and post-intervention assessments measuring HPV knowledge, health beliefs, and vaccination intention. The model allows comparison of outcomes between groups to evaluate the effectiveness of the stage-based educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): TTM-based structured educational program tailored to the participant's stage of readiness for HPV vaccination
  Interventions: Behavioral: TTM-Based Educational Program
- Control Group (No Intervention): No structured education; participants receive no TTM-based training during the study period.

INTERVENTIONS:
Behavioral: TTM-Based Educational Program — A structured, stage-matched educational intervention based on the Transtheoretical Model, delivered face-to-face in five modules aligned with Precontemplation, Contemplation, Preparation, Action, and Maintenance stage
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to examine the impact of a structured educational program based on the Transtheoretical Model (TTM) on HPV knowledge, health beliefs, and vaccination behavioral intentions among first-year nursing students. The study will also evaluate how the intervention affects students' HPV vaccine readiness compared to the TTM.

The primary questions addressed by the study are:

* Does the TTM-based educational intervention increase students' knowledge about HPV and the HPV vaccine?
* Does the program change students' health beliefs regarding susceptibility, severity, benefits, and barriers to HPV and the HPV vaccine?
* Does the program improve students' intentions and readiness to receive the HPV vaccine?
* Do students move to a higher behavioral readiness stage (from Precontemplation to Contemplation, Preparation, Action, or Maintenance) after the intervention?

The researcher will compare the TTM-based educational intervention with a control group that did not receive structured education to determine whether a personalized, stage-based approach is more effective in improving HPV-related outcomes among nursing students.

Participants will:

* Complete baseline questionnaires measuring HPV knowledge, health beliefs, and vaccination intention.
* The experimental group (intervention group) will receive personalized TTM-based education, face-to-face instruction in modules aligned with the five TTM phases (Precontemplation, Contemplation, Preparation, Action, and Maintenance).
* The experimental group will participate in educational sessions designed to raise awareness, correct misinformation, support decision-making, and encourage protective behaviors.
* The control group will not receive any educational program.
* All participants in the experimental and control groups will complete the same questionnaires again to assess changes after the intervention.

The TTM-based educational intervention provides:

* Staged counseling
* Information about HPV and the HPV vaccine
* Activities to raise awareness, strengthen motivation, and support vaccination adoption
* Personalized feedback based on student readiness
* Structured modules focusing on knowledge, belief, and behavior change strategies

The study population included first-year nursing students enrolled in the Faculty of Health Sciences. A total of 88 participants will be recruited and randomly assigned to either the intervention (n=44) or control (n=44) groups through simple randomization.

The results of this study are expected to contribute to the development of evidence-based education strategies in nursing, support of behavioral change models in health education, and strengthen the role of future nurses in HPV prevention, vaccine advocacy, and public health practice.

ELIGIBILITY:
Inclusion Criteria:

* First-year students enrolled in the Nursing Department of the Faculty of Health Sciences
* Provide written informed consent to participate
* Agree to attend all educational sessions and data collection appointments during the study period
* Have sufficient Turkish literacy to read and understand study materials
* Have not previously received any comprehensive education about HPV infection or HPV vaccination

Exclusion Criteria:

* Students who do not agree to participate in the study
* Students who do not provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Vaccination Behavior Intention Scale | Baseline and after completion of the 10-week intervention (5 sessions delivered every 2 weeks)
  Behavioral intention to receive the HPV vaccine will be assessed using the HPV Vaccination Intention Scale, a 6-item instrument developed based on the Theory of Planned Behavior. The scale evaluates participants' intention to receive the HPV vaccine, with higher scores indicating stronger intention to be vaccinated. The secondary outcome is the change in intention score from baseline to post-intervention.

SECONDARY OUTCOMES:
HPV Knowledge Scale | Baseline and after completion of the 10-week intervention (5 sessions delivered every 2 weeks)
  HPV knowledge will be measured using the HPV Knowledge Scale (HPV-BS), a validated 33-item instrument consisting of four subscales: general HPV knowledge (16 items), HPV screening knowledge (6 items), HPV vaccine knowledge (5 items), and HPV vaccination program knowledge (6 items). Total scores range from 0 to 35, with higher scores indicating greater knowledge about HPV infection, transmission, screening, and vaccination. A Cronbach's alpha coefficient of 0.96 was reported in the Turkish validity and reliability study. The primary outcome is the change in total HPV knowledge score from baseline to postintervention.
Health Belief Model Scale regarding HPV and vaccination | Baseline and after completion of the 10-week intervention (5 sessions delivered every 2 weeks)
  Health beliefs regarding HPV and HPV vaccination will be measured using the Health Belief Model Scale (HBM-HPV), a validated instrument developed by Kim (2016) and adapted into Turkish by Guvenc et al. (2016). The scale consists of four subscales: perceived benefits (items 1-3), perceived susceptibility (items 4-5), perceived severity (items 6-9), and perceived barriers (items 10-13 and 15). Higher scores indicate stronger beliefs within each construct. Except for perceived barriers, all subscales are positively associated with HPV vaccination intention. Cronbach's alpha values for the subscales range from 0.71 to 0.78. The secondary outcome is the change in subscale scores from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Adana, CUKUROVA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves identifiable student information, and sharing raw data may pose confidentiality and privacy risks. Data will be stored securely and used only for the purposes approved by the ethics committee. Only aggregated and de-identified results will be reported in publications.